CLINICAL TRIAL: NCT03122574
Title: A Feasibility Study of the Effects of Aromatherapy on the Incidence and Severity of Acute Pain in Pediatric Patients
Brief Title: The Effects of Aromatherapy on the Incidence and Severity of Acute Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: American University (Other)
Responsible Party: Principal Investigator, Katherine Curtin, Clinical Research Coordinator, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro0006362
Record Dates: First submitted 2017-04-03; First posted 2017-04-21 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Venipuncture
Keywords: aromatherapy; pediatric; venipuncture; lavender; pain management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment (Experimental): Pure (100%) lavender aromatherapy
  Interventions: Other: Lavender Aromatherapy
- Placebo Control (Placebo Comparator): Pure (100%) jojoba aromatherapy
  Interventions: Other: Jojoba Aromatherapy
- Standard of care Control (No Intervention): No aromatherapy control group

INTERVENTIONS:
Other: Lavender Aromatherapy — 100% pure lavender aromatherapy was administered using person essential oil diffusor sachets, consisting of three drops of oil on a surgical sponge covered in a sealed plastic packet.
  Arms: Treatment
Other: Jojoba Aromatherapy — 100% pure jojoba aromatherapy was administered using person essential oil diffusor sachets, consisting of three drops of oil on a surgical sponge covered in a sealed plastic packet. This colorless, odorless oil was used as a placebo comparator.
  Arms: Placebo Control

SUMMARY:
The purpose of this research was to estimate feasibility of an aromatherapy pain management intervention to reduce pain and distress caused by venipunctures in a pediatric population. The feasibility of the use of aromatherapy essential oil lavandula angustifolia for pain management intervention (Treatment Group) was compared to placebo aromatherapy with jojoba oil (Placebo Control Group) and to the current standard of care, which is no oil during a venipuncture (Standard of Care Control Group). Primary measured outcomes were assessed using a double-blind randomized design. The physiological measure of heart rate was taken over the course of four minutes at three different intervals to note the pattern of change that occurs during anticipatory anxiety resulting from the impending procedure, the procedural pain experienced during the venipuncture, and the residual fear common after completion of the venipuncture procedure. The Visual Analogue Scale (VAS) for pain and the Hospital Fears Rating Scale (HFRS) were administered to measure subjective pain and anxiety. Participants (N=21) were recruited from the Laboratory Medicine Unit of Children's National Health System. Feasibility was estimated based on the ability to inhale the full dose of oil without adverse effects and and ability to inhale the full dose within the ten-minute time frame. This study analyzed the effect of the aromatherapy pain management intervention, lavandula angustifolia aromatherapy, on the stress response of a pediatric population through observation of physiological and psychological indicators of pain and distress, in order to learn more about the pain and anxiety experienced during venipuncture and the use of aromatherapy to decrease pain and anxiety during venipuncture.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for venipuncture
* English speaking
* Parental written consent
* Child's verbal assent

Exclusion Criteria:

* Essential oil allergy
* Peanut allergy (nut oils processed by manufacturer)
* Medical hypersensitivity to smell
* Asthma triggered by foreign scent
* Frequent venipuncture (5 or more a year)
* Current pain or anxiety medication

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Percentage of participants who complete the intervention in the ten-minute time frame without an adverse event, assessed by stop-watch recording and RN monitoring. | Minute 10
  Adverse event: defined as verbalization of headache, nausea, or dislike of fragrance.

SECONDARY OUTCOMES:
Physiological-heart rate | Minute 3, Minute 5, Minute 7
  Heart rate (raw score) as measured using a NONIN Onyx finger cuff. It took approximately 10 seconds to record. Heart rate was measured (1) two-minutes prior to venipuncture, (2) during venipuncture, and (3) two minutes post-venipuncture, covering in total a 4 minute time span.
Psychological- Visual Analogue Scale (VAS) for pain | Minute 10
  The VAS for pain is a self-report measure that assesses subjective patient pain on a scale from 0-10. It was administered at the end of the 10 minute study and took approximately one minute to administer.
Psychological- Hospital Fears Rating Scale (HFRS) | Minute 1, Minute 10
  The Hospital Fears Rating Scale is a measure of subjective self-report patient anxiety. Scores range from 1-5.It was administered at minute one and again at minute 10 of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine B Curtin, MA, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No